CLINICAL TRIAL: NCT00697359
Title: An Observational Study to Assess the Efficacy of Continuous Subcutaneous Arrhythmia Monitoring Versus Conventional Ambulatory ECG-monitoring in Detecting Atrial Fibrillation in Patients After Pulmonary Vein Isolation
Brief Title: Implantable Loop Recorder Versus Conventional Ambulatory Monitoring in Detecting Atrial Fibrillation After Pulmonary Vein Isolation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Axel Brandes, Associate Professor, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AF-ABL-R-001; S-20080066
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Monitoring; Pulmonary vein isolation; Implantable loop recorder
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): There is only one group in this cohort study.
  Interventions: Device: Implantable loop recorder (ILR)

INTERVENTIONS:
Device: Implantable loop recorder (ILR) — The ILR will be implanted subcutaneous following standard surgical procedure.
  Other Names: All patients in the group get an ILR implanted.

SUMMARY:
The primary aim of the study is to assess the efficacy of continuous rhythm monitoring with an implantable loop recorder (ILR) compared to conventional ambulatory electrocardiography in detecting episodes of atrial fibrillation after pulmonary vein isolation (PVI). The secondary aim is to assess the efficacy of PVI during a two years follow-up and to assess the reliability of the implantable loop recorder in detecting atrial fibrillation.

50 patients will be enrolled into the study. After enrollment an implantable loop recorder will be implanted at least 6 weeks before scheduled PVI. All patients will be followed for 24 months after PVI. During the follow-up period a 72-hours ambulatory electrocardiographic monitoring will be performed at 1, 6, 12, 18, and 24 months. Transthoracic echocardiography will be performed at enrollment, 3, 12, and 24 months after PVI. Moreover, quality of life will be assessed at baseline, and 6 and 12 months after PVI.

ELIGIBILITY:
Inclusion Criteria:

* Age => 30 to =< 70 years
* Documentation of paroxysmal atrial fibrillation
* Documentation of persistent atrial fibrillation of < 3 months duration termination either spontaneously or by DC cardioversion
* Scheduled pulmonary vein isolation
* Treatment with at least one class IC or class III antiarrhythmic drug tried

Exclusion Criteria:

* Atrial fibrillation episodes > 3 months or permanent atrial fibrillation
* No indication for pulmonary vein isolation
* Contraindications for anticoagulation treatment
* No informed consent

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-06; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with atrial fibrillation detected by implantable loop recorder and number of patients with atrial fibrillation detected by conventional ambulatory electrocardiographic monitoring | 12 months

SECONDARY OUTCOMES:
Number of asymptomatic and symptomatic atrial fibrillation episodes | 12 months
Number of symptomatic and asymptomatic atrial fibrillation episodes | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Axel Brandes, MD, Principal Investigator — Odense University Hospital
Locations (3):
- Odense University Hospital, Odense, Denmark
- Academician E. N. Meshalkin, Novosibirsk, Russia
- Örebro University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bjorkenheim A, Brandes A, Magnuson A, Chemnitz A, Edvardsson N, Poci D. Patient-Reported Outcomes in Relation to Continuously Monitored Rhythm Before and During 2 Years After Atrial Fibrillation Ablation Using a Disease-Specific and a Generic Instrument. J Am Heart Assoc. 2018 Feb 24;7(5):e008362. doi: 10.1161/JAHA.117.008362. PMID 29478027
- [Derived] Bjorkenheim A, Brandes A, Chemnitz A, Magnuson A, Edvardsson N, Poci D. Rhythm Control and Its Relation to Symptoms during the First Two Years after Radiofrequency Ablation for Atrial Fibrillation. Pacing Clin Electrophysiol. 2016 Sep;39(9):914-25. doi: 10.1111/pace.12916. Epub 2016 Aug 5. PMID 27418324